CLINICAL TRIAL: NCT00073047
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Multi-center, Dose-ranging Study of Intravenous Daclizumab in Patients With Moderate-to-severe Ulcerative Colitis
Brief Title: Humanized Anti-IL-2 Receptor Monoclonal Antibody in Moderate-to-severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Responsible Party: Nancy Teasdale, Director, Regulatory Affairs
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1008
Record Dates: First submitted 2003-11-14; First posted 2003-11-18 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Ulcerative Colitis; Gastrointestinal Disease; Inflammatory Bowel Disease
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease; Gastrointestinal; Humanized Monoclonal antibody
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Diseases; Inflammatory Bowel Diseases | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
The purpose of The PROSPECT Study is to evaluate an investigational medication for the treatment of moderate to severe ulcerative colitis. This study is being conducted at up to 38 clinical research centers in the US, Canada, and Belgium, and is open to male and female patients 12 years and older. Participants in the study will have a number of visits to a research center over a five-month period. All study related care and medication is provided to qualified participants at no cost: this includes all visits, examinations, and laboratory work.

ELIGIBILITY:
* Moderate to severe active ulcerative colitis diagnosed for at least 4 months.
* Mayo score of 5-10 (inclusive)
* Not used any investigational therapy for 30 days prior to screening
* No treatment with monoclonal antibody therapy within 12 weeks of screening
* No prior treatment with daclizumab

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2003-04; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (30):
  - Clinical Research Associates, Huntsville, Alabama
  - Advanced Medical Research Institute, Anaheim, California
  - Research Foundation of America, Los Angeles, California
  - Western Gastroenterology Group, Los Angeles, California
  - Cedar Sinai Medical Center, Los Angeles, California
  - GVAMC, Gainesville, Florida
  - Clinical Research Associates, Hollywood, Florida
  - Physician Office, Jacksonville, Florida
  - Mount Sinai Medical Center, North Miami Beach, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - The University of Chicago Hospital, Chicago, Illinois
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Drug Research Services, Inc., Metairie, Louisiana
  - Medlantic Investigators Network, Annapolis, Maryland
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Long Island Clinical Research Associates, Great Neck, New York
  - New York Center for Clinical Research, Lake Success, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Columbia Gastro Associates, Columbia, South Carolina
  - Memphis Gastroenterology Group, P.C., Memphis, Tennessee
  - Nashville Medical Research, Nashville, Tennessee
  - Fletcher Allen Health Care, South Burlington, Vermont
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Richmond GI Research Group, Richmond, Virginia
  - McGuire DVAMC, Richmond, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Universitair Ziekenhuis Gasthuisberg, Leuven, Belgium
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Science Center, London, Ontario
  - Montreal General Hospital, Montreal, Quebec

REFERENCES:
- See also: Crohn's and Colitis Foundation of America — http://www.ccfa.org